CLINICAL TRIAL: NCT05091658
Title: Period Tracker Lay User Study
Status: Completed | Type: Observational
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PROTOCOL-1337
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Menstrual Cycles

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: LH Urine Test — Test for qualitative detection of LH in urine

SUMMARY:
This study will assess the ability of the lay user to obtain and record a result. Comprehension of the instructions for use of the product will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18 to 45 years
* Willing to give informed consent and comply with the investigational procedures

Exclusion Criteria:

* Used Clearblue® me Period Tracker app Persona or FAM within the last six months
* Currently or previously employed by SPD, Abbott, Alere, Unipath, P&G or affiliates
* Has an immediate* relative currently or previously (within past 5 years) employed by SPD, Abbott, Alere, Unipath or P&G, or affiliates
* Is a qualified or trainee healthcare professional (HCP)
* Has professional experience of using dipstick type tests or lateral flow devices
* Currently breastfeeding, pregnant or seeking to conceive
* Currently menstruating∆ *Immediate relatives are defined as parents, children, siblings or partner/spouse ∆Volunteer can start the study when their period has ended.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females are representative of the intended user of the product
Study Population: Women between the ages of 18 to 45 represent the intended user of the product
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Lay user usage | 1 hour
  Ability of the lay user to perform a test and record their result

SECONDARY OUTCOMES:
Comprehension of instructions for use | 1 hour
  Ability of the lay user to understand the information provided in the instructions for use

OTHER OUTCOMES:
Lay user ability to read a high and a low result | 1 hour
  Ability of the lay user to score a positive result above a baseline result using the product scoring scale

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Bond, Principal Investigator — SPD Development Company; Raniero Zazzeroni, Study Director — SPD Development Company
Locations (1):
- SPD Development Company Ltd, Bedford, Bedfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data